CLINICAL TRIAL: NCT00357240
Title: Randomized, Open-Label, Multiple-Dose Study to Evaluate the Effect of Omeprazole 20 mg on the Pharmacokinetics of Atazanavir Administered With Ritonavir in Healthy Subjects
Brief Title: Drug Interaction Study With Proton Pump Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AI424-288
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: Protease inhibitor
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; atazanavir, ritonavir drug combination

ARMS (8):
- A1 (Active Comparator)
  Interventions: Drug: Atazanavir
- A2 (Active Comparator)
  Interventions: Drug: Atazanavir/Ritonavir
- A3 I (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir+Omeprazole
- A3 II (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir+Omeprazole
- B1 (Active Comparator)
  Interventions: Drug: Atazanavir
- B2 (Active Comparator)
  Interventions: Drug: Atazanavir/Ritonavir
- B3 I (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir+Omeprazole
- B3 II (Experimental)
  Interventions: Drug: Atazanavir/Ritonavir+Omeprazole

INTERVENTIONS:
Drug: Atazanavir — Capsules, Oral, 400 mg, once daily, 6 days.
  Other Names: Reyataz
  Arms: A1
Drug: Atazanavir/Ritonavir — Capsules/capsules, Oral, 300/100 mg, once daily, 10 days.
  Other Names: Reyataz
  Arms: A2
Drug: Atazanavir/Ritonavir+Omeprazole — Capsules/capsules + Capsules, Oral, 300/100 mg + 20 mg, once daily in PM + once daily in AM, 7 days.
  Other Names: Reyataz
  Arms: A3 I
Drug: Atazanavir/Ritonavir+Omeprazole — Capsules/capsules + Capsules, Oral, 400/100 mg + 20 mg, once daily in PM + once daily in AM, 7 days.
  Other Names: Reyataz
  Arms: A3 II
Drug: Atazanavir — Capsules, Oral, 400 mg, once daily, 6 days.
  Other Names: Reyataz
  Arms: B1
Drug: Atazanavir/Ritonavir — Capsules/capsules, Oral, 300/100 mg, once daily, 10 days.
  Other Names: Reyataz
  Arms: B2
Drug: Atazanavir/Ritonavir+Omeprazole — Capsules/capsules + Capsules, Oral, 400/100 mg + 20 mg, once daily in AM + once daily in AM, 7 days.
  Other Names: Reyataz
  Arms: B3 I
Drug: Atazanavir/Ritonavir+Omeprazole — Capsules/capsules + Capsules, Oral, 400/100 mg + 20 mg, once daily in AM + once daily in PM, 7 days.
  Other Names: Reyataz
  Arms: B3 II

SUMMARY:
The purpose of this clinical research study is to assess the effect of omeprazole at 20 mg on the pharmacokinetics of atazanavir administered as atazanavir with ritonavir relative to atazanavir or atazanavir/ritonavir in the absence of omeprazole in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 to 50 years old with BMI 18 to 32 kg/m2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Effect of omeprazole 20 mg on PK of atazanavir (with ritonavir), coadministered or temporally separated, in healthy subjects.

SECONDARY OUTCOMES:
PK of ritonavir and omeprazole. Safety and tolerability of atazanavir +/- ritonavir, +/- omeprazole.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hamilton, New Jersey, United States